CLINICAL TRIAL: NCT06732869
Title: PACE - Physical Activity in COPD Using E-Health: Effectiveness of a Personalised eHealth Platform Integrated Into Pulmonary Rehabilitation to Increase Physical Activity in Patients With COPD - a Randomized Controlled Trial
Brief Title: Effectiveness of a Physical ACtivity Coaching Intervention Using E-Health for COPD Patients in Pulmonary Rehabilitation
Acronym: PACE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Instituto Politécnico de Leiria (Other)
Collaborators: Unidade Local de Saúde do Baixo Mondego (Unknown); Unidade Local de Saúde de Lisboa Norte (Unknown); Faculdade de Motricidade Humana de Lisboa (Unknown)
Responsible Party: Principal Investigator, Sofia Flora, Principal Investigator, Instituto Politécnico de Leiria
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ciTechCare_PhD_SF; doi.org/10.54499/2020.06954.BD (Other Grant/Funding Number: Foundation for Science and Technology (FCT)); UIDB/05704/2020 (Other Grant/Funding Number: ciTechCare, Polytechnic of Leiria)
Record Dates: First submitted 2024-11-27; First posted 2024-12-13 (Actual); Last update posted 2024-12-13 (Actual); Status verified 2024-12

CONDITIONS: COPD; Physical Activity
Keywords: physical activity; COPD; eHealth; pulmonary rehabilitation
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Motor Activity

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental Group - Pulmonary rehabilitation + eHealth physical activity coaching intervention (Experimental): Patients will attend a PR program for 10 weeks and receive an eHealth PA coaching intervention (smartband connected to a mobile application) in the week 5 of PR until months after end of PR.
  Interventions: Behavioral: eHealth physical activity coaching intervention; Behavioral: pulmonary rehabilitation
- Control group - pulmonary rehabilitation (Other): Patients will attend pulmonary rehabilitation program for 10 weeks.
  Interventions: Behavioral: pulmonary rehabilitation

INTERVENTIONS:
Behavioral: eHealth physical activity coaching intervention — Patients will attend a PR program and in week 5 of PR will receive an eHealth PA coaching intervention until 6 months after end of PR. The PA goals will be prescribed through a phone call and the personalisation of goal prescription will be based on an algorithm considering patient's performance in the previous week, perceived easiness of achieving the previous goal and confidence to change it. If patient does not achieve the goal, reasons, barriers to PA and strategies to overcome them will be identified. Patients will receive a daily notification about their goal achievements, at 6PM every day, giving them the possibility to increase their PA to achieve the goal, if they have not reached it yet. Patients will also receive personalized notifications sent manually by the researcher whenever appropriate. PA goals will be prescribed on a weekly basis.
  Arms: Experimental Group - Pulmonary rehabilitation + eHealth physical activity coaching intervention
Behavioral: pulmonary rehabilitation — Patients will attend pulmonary rehabilitation program for 10 weeks. Pulmonary rehabilitation is evidence-based multidisciplinary intervention based on thorough patient assessment followed by patient-tailored therapies that include, but are not limited to exercise training, education, self-management intervention aiming at behaviour change, known to improve health status and psychological well-being, reducing dyspnoea and healthcare utilization and hospitalization. In this study, pulmonary rehabilitation programs will have 20 sessions, twice a week, including exercise training (aerobic and strength training), educational sessions about topics as medication, smoking cessation, energy conservation techniques, physical activity, stress and anxiety management, breathing control, inhaled therapy and nutrition; nutritional and psychosocial counselling. Education session about PA importance and recommendations will be also provided in both arms.

SUMMARY:
The goal of this randomized controlled trial is to evaluate the efficacy of a physical activity coaching intervention - delivered through an eHealth platform both during and after pulmonary rehabilitation - to enhance physical activity levels and health-related outcomes in patients with Chronic Obstructive Pulmonary Disease (COPD). All participants will attend the pulmonary rehabilitation program for 2 months; the experimental group will receive a physical activity coaching intervention at the end of the 1st month of the rehabilitation program, which will continue for 6 months following the completion of the program. Assessments will be conducted at the beginning, midway, and at the end of the coaching program, as well as 3 months and 6 months after its conclusion.

DETAILED DESCRIPTION:
This randomized controlled trial aims to evaluate the efficacy of a physical activity coaching intervention - delivered through an eHealth platform, both during and after pulmonary rehabilitation - to enhance physical activity levels and health-related outcomes in patients with Chronic Obstructive Pulmonary Disease (COPD).

All participants will attend the pulmonary rehabilitation program for 10 weeks. At week 5 of the rehabilitation program, the experimental group will receive a physical activity coaching intervention, which will continue for 6 months following its completion. This intervention will include an eHealth platform divided into two applications (a mobile app for patients and a web app for researchers/healthcare professionals).

Goal setting and progression according to patients' performance and willingness to increase will occur every week, through phone calls. Barriers to physical activity and strategies to overcome them will be identified between the patient and researcher, during the goal-setting moments. Notifications about PA goals achievement and incentives will be sent to patients during the intervention.

The assessment moments will be conducted at the beginning, midway, and end of the pulmonary rehabilitation program, as well as 3- and 6 months after its conclusion.

ELIGIBILITY:
Inclusion criteria:

* age > 40 years old
* diagnosis of COPD according to GOLD criteria, clinically stable (i.e., with no exacerbations in the previous month)
* being enrolled in a pulmonary rehabilitation program
* having a smartphone with access to the internet
* being able to understand and provide informed consent.

Exclusion criteria:

* simultaneous participation in another behavioural modification program
* having any clinical condition that precludes participation in a PA intervention (e.g., severe musculoskeletal or neurological disorders and unstable cardiovascular disease)
* another primary respiratory disease
* history of recent neoplasia (including last treatment) in the previous year.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 57 (Estimated)
Dates: Start 2024-12-02 (Actual); Primary Completion 2025-06 (Estimated); Study Completion 2025-06 (Estimated)

PRIMARY OUTCOMES:
Accelerometry (number of daily steps) | weeks 1, 5, 10 of pulmonary rehabilitation program and 3- and 6-months after its conclusion
  PA will be objectively measured using the triaxial accelerometer Actigraph GT3X+, already validated in COPD. Patients will be instructed to wear the accelerometer for 7 days on the dominant side of their waist, held by an elastic strap, during waking hours, except for bathing or swimming. A valid day will be defined as a minimum of 8 hours of wearing time, and patients will need to have at least 4 valid days in each moment of data collection. Accelerometer-based data will be then downloaded and analysed using the algorithms of Freedson (1998) with 60-s epoch: daily time (in min) spent in light-intensity PA, moderate, vigorous and a combination of both. The number of steps per day and per week will also be collected, being the main outcome of the study.

SECONDARY OUTCOMES:
6-Minute Walk Test (exercise capacity) | weeks 1, 5, 10 of pulmonary rehabilitation program and 3- and 6-months after its conclusion
  Functional exercise capacity was measured using 6MWT, and predicted values were computed using the equation developed for Portuguese adults. The test will be conducted according to guidelines from ERS/ATS.
modified Medical Research Council (Dyspnoea) | weeks 1, 5, 10 of pulmonary rehabilitation program and 3- and 6-months after its conclusion
  Dyspnoea was assessed through the modified Medical Research Council (mMRC), on a scale from 0 to 4, in which 0 means 'dyspnoea only with strenuous exercise' and 4 means 'too dyspnoeic to leave house or breathless when dressing'.
Checklist of Individual Strength (Fatigue) | weeks 1, 5, 10 of pulmonary rehabilitation program and 3- and 6-months after its conclusion
  Fatigue will be assessed with the Checklist of Individual Strength (CIS20). This questionnaire consists of four dimensions (Subjective Fatigue, Concentration, Motivation and Physical Activity) that assess the fatigue severity.
COPD Assessment Test (Impact of symptoms on health status) | weeks 1, 5, 10 of pulmonary rehabilitation program and 3- and 6-months after its conclusion
  The COPD Assessment Test is designed to measure the impact of COPD on a person's life, and how this changes over time.The total score is a sum of the 8 questions. Higher scores indicates worse impact of the disease.
MOS Short-Form Health Survey 36 Item v2 (SF-36) (Quality of Life) | weeks 1, 5, 10 of pulmonary rehabilitation program and 3- and 6-months after its conclusion
  Quality of Life will be assessed with MOS Short-Form Health Survey 36 Item v2 (SF-36). The SF-36 is widely used to measure perceived health-related quality of life. The instrument includes scales for physical functioning, social functioning, limitations in function due to physical or emotional problems, mental health, energy, pain and general perception of health. The score ranges from 0 - 100 (higher scores indicate better levels of quality of life.
Physical Exercise Self-Efficacy Scale (self-efficacy for PA) | weeks 1, 5, 10 of pulmonary rehabilitation program and 3- and 6-months after its conclusion
  self-efficacy for PA will be assessed with Physical Exercise Self-Efficacy Scale which consists of 5 items that analyse an individual's confidence in performing physical exercise according to different emotional states (worried, depressed, nervous, tired and busy). The total score is the sum of the scores for each item, ranging from 5 to 20. The higher the score, the greater the belief or sense of self-efficacy for exercise.

CONTACTS AND LOCATIONS:
Overall Officials: Sofia Flora, PT, MSc, Principal Investigator — Center for Innovative Care and Health Technology, Polytechnic of Leiria
Locations (1):
- Center for Innovative Care and Health Technology (ciTechCare), Polytechnic of Leiria, Leiria, Portugal

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Global Strategy for the Diagnosis Management and Prevention of COPD, Global Initiative for Chronic Obstructive Lung Disease (GOLD). Available from: https://goldcopd.org/2024-gold-report/. 2024.
- [Background] McCarthy B, Casey D, Devane D, Murphy K, Murphy E, Lacasse Y. Pulmonary rehabilitation for chronic obstructive pulmonary disease. Cochrane Database Syst Rev. 2015 Feb 23;2015(2):CD003793. doi: 10.1002/14651858.CD003793.pub3. PMID 25705944
- [Background] Ding D, Lawson KD, Kolbe-Alexander TL, Finkelstein EA, Katzmarzyk PT, van Mechelen W, Pratt M; Lancet Physical Activity Series 2 Executive Committee. The economic burden of physical inactivity: a global analysis of major non-communicable diseases. Lancet. 2016 Sep 24;388(10051):1311-24. doi: 10.1016/S0140-6736(16)30383-X. Epub 2016 Jul 28. PMID 27475266
- [Background] Puhan MA, Gimeno-Santos E, Cates CJ, Troosters T. Pulmonary rehabilitation following exacerbations of chronic obstructive pulmonary disease. Cochrane Database Syst Rev. 2016 Dec 8;12(12):CD005305. doi: 10.1002/14651858.CD005305.pub4. PMID 27930803
- [Background] Spruit MA, Singh SJ, Garvey C, ZuWallack R, Nici L, Rochester C, Hill K, Holland AE, Lareau SC, Man WD, Pitta F, Sewell L, Raskin J, Bourbeau J, Crouch R, Franssen FM, Casaburi R, Vercoulen JH, Vogiatzis I, Gosselink R, Clini EM, Effing TW, Maltais F, van der Palen J, Troosters T, Janssen DJ, Collins E, Garcia-Aymerich J, Brooks D, Fahy BF, Puhan MA, Hoogendoorn M, Garrod R, Schols AM, Carlin B, Benzo R, Meek P, Morgan M, Rutten-van Molken MP, Ries AL, Make B, Goldstein RS, Dowson CA, Brozek JL, Donner CF, Wouters EF; ATS/ERS Task Force on Pulmonary Rehabilitation. An official American Thoracic Society/European Respiratory Society statement: key concepts and advances in pulmonary rehabilitation. Am J Respir Crit Care Med. 2013 Oct 15;188(8):e13-64. doi: 10.1164/rccm.201309-1634ST. PMID 24127811
- [Background] Spruit MA, Pitta F, McAuley E, ZuWallack RL, Nici L. Pulmonary Rehabilitation and Physical Activity in Patients with Chronic Obstructive Pulmonary Disease. Am J Respir Crit Care Med. 2015 Oct 15;192(8):924-33. doi: 10.1164/rccm.201505-0929CI. PMID 26161676
- [Background] Burge AT, Cox NS, Abramson MJ, Holland AE. Interventions for promoting physical activity in people with chronic obstructive pulmonary disease (COPD). Cochrane Database Syst Rev. 2020 Apr 16;4(4):CD012626. doi: 10.1002/14651858.CD012626.pub2. PMID 32297320
- [Background] Wilson JJ, O'Neill B, Collins EG, Bradley J. Interventions to Increase Physical Activity in Patients with COPD: A Comprehensive Review. COPD. 2015 Jun;12(3):332-43. doi: 10.3109/15412555.2014.948992. Epub 2014 Sep 15. PMID 25221907
- [Background] Jiang X, Ming WK, You JH. The Cost-Effectiveness of Digital Health Interventions on the Management of Cardiovascular Diseases: Systematic Review. J Med Internet Res. 2019 Jun 17;21(6):e13166. doi: 10.2196/13166. PMID 31210136
- [Background] Kowatsch, T., et al., Design and Evaluation of a Mobile Chat App for the Open Source Behavioral Health Intervention Platform MobileCoach. 2017. 485-489
- [Background] Blazun H, Saranto K, Kokol P, Vosner J. Information and communication technology as a tool for improving physical and social activity of the elderly. NI 2012 (2012). 2012 Jun 23;2012:26. eCollection 2012. PMID 24199042
- [Background] Solanas, A., et al., Smart health: A context-aware health paradigm within smart cities. IEEE Communications Magazine, 2014. 52(8): p. 74-81.
- [Background] Laranjo L, Ding D, Heleno B, Kocaballi B, Quiroz JC, Tong HL, Chahwan B, Neves AL, Gabarron E, Dao KP, Rodrigues D, Neves GC, Antunes ML, Coiera E, Bates DW. Do smartphone applications and activity trackers increase physical activity in adults? Systematic review, meta-analysis and metaregression. Br J Sports Med. 2021 Apr;55(8):422-432. doi: 10.1136/bjsports-2020-102892. Epub 2020 Dec 21. PMID 33355160
- [Background] Sim I. Mobile Devices and Health. N Engl J Med. 2019 Sep 5;381(10):956-968. doi: 10.1056/NEJMra1806949. No abstract available. PMID 31483966
- [Background] Demeyer H, Louvaris Z, Frei A, Rabinovich RA, de Jong C, Gimeno-Santos E, Loeckx M, Buttery SC, Rubio N, Van der Molen T, Hopkinson NS, Vogiatzis I, Puhan MA, Garcia-Aymerich J, Polkey MI, Troosters T; Mr Papp PROactive study group and the PROactive consortium. Physical activity is increased by a 12-week semiautomated telecoaching programme in patients with COPD: a multicentre randomised controlled trial. Thorax. 2017 May;72(5):415-423. doi: 10.1136/thoraxjnl-2016-209026. Epub 2017 Jan 30. PMID 28137918
- [Background] Boutron I, Altman DG, Moher D, Schulz KF, Ravaud P; CONSORT NPT Group. CONSORT Statement for Randomized Trials of Nonpharmacologic Treatments: A 2017 Update and a CONSORT Extension for Nonpharmacologic Trial Abstracts. Ann Intern Med. 2017 Jul 4;167(1):40-47. doi: 10.7326/M17-0046. Epub 2017 Jun 20. PMID 28630973
- [Background] Eysenbach G; CONSORT-EHEALTH Group. CONSORT-EHEALTH: improving and standardizing evaluation reports of Web-based and mobile health interventions. J Med Internet Res. 2011 Dec 31;13(4):e126. doi: 10.2196/jmir.1923. PMID 22209829
- [Background] Faul F, Erdfelder E, Lang AG, Buchner A. G*Power 3: a flexible statistical power analysis program for the social, behavioral, and biomedical sciences. Behav Res Methods. 2007 May;39(2):175-91. doi: 10.3758/bf03193146. PMID 17695343
- [Background] Demeyer H, Burtin C, Hornikx M, Camillo CA, Van Remoortel H, Langer D, Janssens W, Troosters T. The Minimal Important Difference in Physical Activity in Patients with COPD. PLoS One. 2016 Apr 28;11(4):e0154587. doi: 10.1371/journal.pone.0154587. eCollection 2016. PMID 27124297
- [Background] Pimenta S, Silva CG, Flora S, Hipolito N, Burtin C, Oliveira A, Morais N, Brites-Pereira M, Carreira BP, Januario F, Andrade L, Martins V, Rodrigues F, Brooks D, Marques A, Cruz J. What Motivates Patients with COPD to Be Physically Active? A Cross-Sectional Study. J Clin Med. 2021 Nov 29;10(23):5631. doi: 10.3390/jcm10235631. PMID 34884333
- [Background] Vorrink SN, Kort HS, Troosters T, Zanen P, Lammers JJ. Efficacy of an mHealth intervention to stimulate physical activity in COPD patients after pulmonary rehabilitation. Eur Respir J. 2016 Oct;48(4):1019-1029. doi: 10.1183/13993003.00083-2016. Epub 2016 Sep 1. PMID 27587557
- [Background] Rochester CL, Vogiatzis I, Holland AE, Lareau SC, Marciniuk DD, Puhan MA, Spruit MA, Masefield S, Casaburi R, Clini EM, Crouch R, Garcia-Aymerich J, Garvey C, Goldstein RS, Hill K, Morgan M, Nici L, Pitta F, Ries AL, Singh SJ, Troosters T, Wijkstra PJ, Yawn BP, ZuWallack RL; ATS/ERS Task Force on Policy in Pulmonary Rehabilitation. An Official American Thoracic Society/European Respiratory Society Policy Statement: Enhancing Implementation, Use, and Delivery of Pulmonary Rehabilitation. Am J Respir Crit Care Med. 2015 Dec 1;192(11):1373-86. doi: 10.1164/rccm.201510-1966ST. PMID 26623686
- [Background] Orchard JW. Prescribing and dosing exercise in primary care. Aust J Gen Pract. 2020 Apr;49(4):182-186. doi: 10.31128/AJGP-10-19-5110. PMID 32233343
- [Background] ZuWallack, C.B.R., Exercise Training in Pulmonary Rehabilitation, in Textbook of Pulmonary Rehabilitation, A.E.H. Enrico Clini, Fabio Pitta, Thierry Troosters, Editor. 2018, Springer Cham
- [Background] Watz H, Pitta F, Rochester CL, Garcia-Aymerich J, ZuWallack R, Troosters T, Vaes AW, Puhan MA, Jehn M, Polkey MI, Vogiatzis I, Clini EM, Toth M, Gimeno-Santos E, Waschki B, Esteban C, Hayot M, Casaburi R, Porszasz J, McAuley E, Singh SJ, Langer D, Wouters EF, Magnussen H, Spruit MA. An official European Respiratory Society statement on physical activity in COPD. Eur Respir J. 2014 Dec;44(6):1521-37. doi: 10.1183/09031936.00046814. Epub 2014 Oct 30. PMID 25359358
- [Background] Michie S, Richardson M, Johnston M, Abraham C, Francis J, Hardeman W, Eccles MP, Cane J, Wood CE. The behavior change technique taxonomy (v1) of 93 hierarchically clustered techniques: building an international consensus for the reporting of behavior change interventions. Ann Behav Med. 2013 Aug;46(1):81-95. doi: 10.1007/s12160-013-9486-6. PMID 23512568
- [Background] Rabinovich RA, Louvaris Z, Raste Y, Langer D, Van Remoortel H, Giavedoni S, Burtin C, Regueiro EM, Vogiatzis I, Hopkinson NS, Polkey MI, Wilson FJ, Macnee W, Westerterp KR, Troosters T; PROactive Consortium. Validity of physical activity monitors during daily life in patients with COPD. Eur Respir J. 2013 Nov;42(5):1205-15. doi: 10.1183/09031936.00134312. Epub 2013 Feb 8. PMID 23397303
- [Background] Demeyer H, Burtin C, Van Remoortel H, Hornikx M, Langer D, Decramer M, Gosselink R, Janssens W, Troosters T. Standardizing the analysis of physical activity in patients with COPD following a pulmonary rehabilitation program. Chest. 2014 Aug;146(2):318-327. doi: 10.1378/chest.13-1968. PMID 24603844
- [Background] Freedson PS, Melanson E, Sirard J. Calibration of the Computer Science and Applications, Inc. accelerometer. Med Sci Sports Exerc. 1998 May;30(5):777-81. doi: 10.1097/00005768-199805000-00021. PMID 9588623
- [Background] Holland AE, Spruit MA, Troosters T, Puhan MA, Pepin V, Saey D, McCormack MC, Carlin BW, Sciurba FC, Pitta F, Wanger J, MacIntyre N, Kaminsky DA, Culver BH, Revill SM, Hernandes NA, Andrianopoulos V, Camillo CA, Mitchell KE, Lee AL, Hill CJ, Singh SJ. An official European Respiratory Society/American Thoracic Society technical standard: field walking tests in chronic respiratory disease. Eur Respir J. 2014 Dec;44(6):1428-46. doi: 10.1183/09031936.00150314. Epub 2014 Oct 30. PMID 25359355
- [Background] Marques A, Rebelo P, Paixao C, Almeida S, Jacome C, Cruz J, Oliveira A. Enhancing the assessment of cardiorespiratory fitness using field tests. Physiotherapy. 2020 Dec;109:54-64. doi: 10.1016/j.physio.2019.06.003. Epub 2019 Jun 18. PMID 32173042
- [Background] ATS Committee on Proficiency Standards for Clinical Pulmonary Function Laboratories. ATS statement: guidelines for the six-minute walk test. Am J Respir Crit Care Med. 2002 Jul 1;166(1):111-7. doi: 10.1164/ajrccm.166.1.at1102. No abstract available. PMID 12091180
- [Background] Agarwala P, Salzman SH. Six-Minute Walk Test: Clinical Role, Technique, Coding, and Reimbursement. Chest. 2020 Mar;157(3):603-611. doi: 10.1016/j.chest.2019.10.014. Epub 2019 Nov 2. PMID 31689414
- [Background] Borg, G., Borg's perceived exertion and pain scales. 1998, Champaign, IL, US: Human Kinetics. viii, 104.
- [Background] Doherty, D.E., et al., Chronic Obstructive Pulmonary Disease: Consensus Recommendations for Early Diagnosis and Treatment. J Fam Pract, 2006. Supplement: p. S1-S8.
- [Background] Vercoulen JH, Swanink CM, Fennis JF, Galama JM, van der Meer JW, Bleijenberg G. Dimensional assessment of chronic fatigue syndrome. J Psychosom Res. 1994 Jul;38(5):383-92. doi: 10.1016/0022-3999(94)90099-x. PMID 7965927
- [Background] Jones PW, Harding G, Berry P, Wiklund I, Chen WH, Kline Leidy N. Development and first validation of the COPD Assessment Test. Eur Respir J. 2009 Sep;34(3):648-54. doi: 10.1183/09031936.00102509. PMID 19720809
- [Background] Ferreira PL. [Development of the Portuguese version of MOS SF-36. Part II --Validation tests]. Acta Med Port. 2000 May-Jun;13(3):119-27. Portuguese. PMID 11026151
- [Background] Ware JE Jr, Sherbourne CD. The MOS 36-item short-form health survey (SF-36). I. Conceptual framework and item selection. Med Care. 1992 Jun;30(6):473-83. PMID 1593914
- [Background] Schwarzer, R. and B. Renner, Health-Specific Self-Efficacy Scales. 2009.
- [Background] Spieth PM, Kubasch AS, Penzlin AI, Illigens BM, Barlinn K, Siepmann T. Randomized controlled trials - a matter of design. Neuropsychiatr Dis Treat. 2016 Jun 10;12:1341-9. doi: 10.2147/NDT.S101938. eCollection 2016. PMID 27354804

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2024-12-04): https://cdn.clinicaltrials.gov/large-docs/69/NCT06732869/Prot_SAP_000.pdf
  • Informed Consent Form (2024-12-04): https://cdn.clinicaltrials.gov/large-docs/69/NCT06732869/ICF_001.pdf